CLINICAL TRIAL: NCT05151874
Title: Valuation of the Evolution of Passive Mobility (ROM)in the Spastic Upper Limb After Injection of Abobotulinumtoxin(Dysport®) in Patients With Post-stroke Spasticity
Brief Title: Valuation of the Evolution of Passive Mobility in the Spastic Upper Limb After Injection of Abobotulinumtoxin(Dysport®)
Acronym: ROM-ICTUS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-ROM-2020-135
Record Dates: First submitted 2021-08-06; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Spasticity, Muscle; Stroke Sequelae; Movement Disorders
Keywords: Spasticity; Abobotulinum toxin; Injection; Rehabilitation
MeSH Terms: conditions — Muscle Spasticity; Movement Disorders | interventions — abobotulinumtoxinA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Range of movement: Change in passive joint mobility (ROM) of the carpus (flexion-extension) affected by spasticity pattern III during a 20-week follow-up.
  Interventions: Drug: Abobotulinum toxin A

INTERVENTIONS:
Drug: Abobotulinum toxin A — To measure ROM evolution in patients with post-stroke spasticity in the upper limb with spasticity pattern III.
  Other Names: toxin infiltration

SUMMARY:
Assessing the objective measurement of passive joint mobility (ROM) in the spastic upper limb with Jost's pattern III in patients with post-stroke spasticity after infiltration with BoNT-A allows to objectify the increase in passive joint balance (ROM).

DETAILED DESCRIPTION:
Changes in joint mobility in patients with post-stroke upper limb spasticity after infiltration of botulinum toxin type A.

The spasticity pattern that will be evaluated will be pattern number III based on the classification of Jost et al. Joint mobility will be measured with the Lynx instrument (DyCare)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years.
* Hemiplegic patients with post-stroke upper limb spasticity affected by pattern III1 who have undergone at least 2 cycles of previous treatment with BoNT-A
* Patients with a MAS scale (Modified Ashworth Scale) between 2 and 3 for the affected muscle group; shoulder, elbow, carpus and metacarpophalangeal.
* Patients with Hackett ultrasound qualitative scale between 2 and 3 for the affected muscle group; shoulder, elbow, carpus and metacarpophalangeal.

Exclusion Criteria:

* Patients who do not wish to sign the informed consent.
* Prior lack of primary or secondary response to any BoNT-A for any specific condition or known sensitivity to BoNT-A or any excipient.
* Routine or prescribed treatment with any medication that directly or indirectly interferes with neuromuscular function in the last 3 months prior to study botulinum toxin treatment.
* Having undergone surgery on the muscles, ligaments, tendons, nerves or bones of the limb to be treated.
* Any medical condition or analytical finding that, in the opinion of the investigator, may compromise compliance with the objectives and / or procedures of the study protocol or exclude the administration of BoNT-A.
* Treatment with an investigational new drug in the 4 weeks or 5 half-lives prior to screening to enter the study.
* Pregnancy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged ≥ 18 years.
  Hemiplegic patients with post-stroke upper limb spasticity affected by pattern III1 who have undergone at least 2 cycles of previous treatment with BoNT-A
  Patients with a MAS scale (Modified Ashworth Scale) between 2 and 3 for the affected muscle group; shoulder, elbow, carpus and metacarpophalangeal.
  Patients with Hackett ultrasound qualitative scale between 2 and 3 for the affected muscle group; shoulder, elbow, carpus and metacarpophalangeal.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in passive range of motion | Through study completion, an average of 1 year
  Change in passive joint mobility (ROM) of the upper limb affected by spasticity pattern III a 20-week follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain